CLINICAL TRIAL: NCT05922384
Title: Safety and Efficacy Study of KL-7SHRNA Injection Solution in the Treatment of AIDS Patients With Lymphoma
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Affiliated Hospital of Guangdong Medical University (Other)
Responsible Party: Principal Investigator, Jinqi Huang, Director of Hematology Department, Affiliated Hospital of Guangdong Medical University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KL210515
Record Dates: First submitted 2023-06-16; First posted 2023-06-28 (Actual); Last update posted 2023-06-28 (Actual); Status verified 2023-06

CONDITIONS: HIV Infections; Lymphoma
Keywords: HIV-1 infection; Lymphoma; gene therapy; 7shRNA
MeSH Terms: conditions — HIV Infections; Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 7shRNA modified CD34+stem cells (Experimental): Patients undergo high-dose chemotherapy or chemoradiotherapy according to institutional guidelines and then received hematopoietic stem cell transplant on day 0
  Interventions: Drug: KL-7SHRNA injection solution

INTERVENTIONS:
Drug: KL-7SHRNA injection solution — Patients continue to receive HAART throughout treatment until meet the criteria of interruption of HAART.
  Other Names: Drug: carmustine Given IV Other Names: BCNU BiCNU bis-chloronitrosourea; Drug: etoposide Given IV Other Names: EPEG VP-16 VP-16-213; Drug: cytosine arabinoside Given IV; Drug: melphalan Given IV

SUMMARY:
This pilot clinical trial studies gene therapy in treating patients with HIV-1 infecetion combined with lymphoma undergoing 7shRNA lentiviral vector transduced CD34+ hematopoietic stem cell transplant. Giving chemotherapy before a stem cell transplant stops the growth of cancer cells by stopping them from dividing or killing them. After treatment, CD34+hematopoietic stem cells are mobilized and collected from the patient's peripheral blood. The CD34+stem cells are then isolated and transduced with lenti-7shRNA vector and reinfused to the patient to replace the blood-forming cells that were destroyed by the chemotherapy.

DETAILED DESCRIPTION:
Primary objectives:

1. To determine the safety and feasibility of using lenti-7shRNA transduced hematopoietic stem/progenitor cells in the setting of autologous hematopoietic cell transplantation for treatment of HIV infection combined with lymphoma. The safety of the genetically modified product used in the transplant procedure will be assessed by monitoring each subject for adverse events (procedure related toxicity); absolute neutrophil count (ANC)/platelet engraftment (sustained recovery); and evidence of replication competent vector or vector recombination with the human immunodeficiency virus (HIV) quasi-species present in the patient.
2. To determine the quantity and duration of vector-marked peripheral blood cells and to characterize: the duration and level of gene marking and expression of the anti-HIV shRNA in these transduced cells, and the characterization of the integration sites of vector sequences in circulating cells if there is a clinical syndrome suggestive of a clonal expansion of hematopoietic cells. In addition, the feasibility of the process will be assessed based on the results of the release testing of the transduced cells prior to injection into the patient.
3. To measure the effect of HIV infection on the presence of HIV-resistant blood cells as measured by genetic marking for vector sequences before and after antiviral treatment interruption.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) 18-25, body weight should be ≥ 40kg;
* Meet the Diagnostic Criteria for AIDS and HIV Infection (WS293-2019), and be diagnosed as HIV seropositive;
* HIV infection combined with lymphoma, in partial remission or relapsed after initial complete remission, failed induction therapy, but responds to salvage therapy;
* Age-adjusted IPI 2-3 points;
* Meet the indications for autologous bone marrow transplantation after clinical evaluation;
* HIV viral load <1000 copies/ml;
* Must have the ability to understand and the willingness to sign a written informed consent.

Exclusion Criteria:

* Any HIV-related uncontrolled opportunistic infection, including fungal infection, sepsis, active tuberculosis, weightlessness, severe diarrhea, active opportunistic infections in the central nervous system or active hepatitis B, hepatitis C, and other viral infections such as CMV;
* Cardiac insufficiency (LVEF<50%), renal insufficiency (creatinine>2mg/dl), hepatic insufficiency (AST/ALT>3 ULN and/or PT <70% unrelated to lymphoma);
* HAART treatment failure (including at least one NRTI, one NNRTI and two PI) and/or CD4 count < 50/cmm);
* Malignancy other than lymphoma, unless (1) in complete remission and more than 5 years from last treatment, or (2) cervical/anal squamous cell carcinoma in situ or (3) superficial basal cell and squamous cell cancers of the skin;
* Participation of other investigational agents (traditional Chinese medicine is not included) within 3 months；
* Any concurrent or past medical condition that, in the opinion of the Investigator, would exclude the subject from participation or any psychosocial conditions that would hinder study compliance or follow-up, at the discretion of the Investigator.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 3 (Estimated)
Dates: Start 2023-07-05 (Estimated); Primary Completion 2025-09-10 (Estimated); Study Completion 2026-04-10 (Estimated)

PRIMARY OUTCOMES:
Overall survival | D0 post-infusion to completion of follow-up, an average of 2 year
  Number of patients alive all over the trial
Engraftment time of 7shRNA modified CD34+ stem cells | within day +28 after gene therapy
  Haematological engraftment is defined as first day of neutrophil count >500/mm3 and platelets >20,000/mm3 on 7 consecutive blood counts.

SECONDARY OUTCOMES:
7shRNA VCN | At week 2, months 1, 2, 3, 4, 5, 6, 7, 8, 9，10,12，15,18,21and 24 post-transplant
  Detection of 7shRNA VCN in CD4+T cells via qPRC.
Duration of interruption of HAART | Up to 24 months post-treatment
  At two months post-transplant, or later, HAART will be voluntarily interrupted only for participants who have a CD4 count of 200 or higher with no detectable viral load and 7shRNA VCN>0.5, for participants in which the CD4 T-cell count has not risen to ≥ 200 cells/mm3 at the time of the planned HAART interruption, HAART will continue until the T-cell count has risen to ≥ 200 cells/mm3.
Transplantation related mortality | Up to 24 months post-treatment
  Number of patients die of transplantation all over the trial

CONTACTS AND LOCATIONS:
Overall Officials: yuming Zhang, PhD, Principal Investigator — Affiliated hospital of Guangdong medical university, Guangdong province, China
Locations (1):
- Affiliated hospital of Guangdong medical university, Zhanjiang, Guangdong, China

IPD SHARING:
Plan to Share IPD: No